CLINICAL TRIAL: NCT00993954
Title: Reduction of Radial Head Subluxation in Children Via a Nurse Initiated Pathway: A Randomized Control Trial
Brief Title: Nurse Reduction of Pulled Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Andrew Dixon, Assistant Professor, University of Alberta
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08/29x
Record Dates: First submitted 2009-10-08; First posted 2009-10-14 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Radial Head Subluxation
Keywords: Nurse Treatment; Pulled Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse Reduction (Experimental): Patients randomized to reduction by nurse.
  Interventions: Procedure: Reduction of Radial Head Subluxation
- Physician Reduction (Active Comparator): Patients randomized to treatment by Emergency Department Physician in traditional ED manner
  Interventions: Procedure: Reduction of Radial Head Subluxation

INTERVENTIONS:
Procedure: Reduction of Radial Head Subluxation — Nurse group will use hyperpronation with extension for first attempt and supination and flexion for second attempt. Physician controls will use either method at their discretion

SUMMARY:
Radial head subluxation, also known as pulled elbow or nursemaid's elbow, is one of the most common upper extremity injuries in young children and a common reason for an emergency department visit.1 The injury typically occurs when a forceful longitudinal traction is applied to an extended and pronated forearm.2 Children with radial head subluxation are usually easily recognized by their clinical presentation and rapidly treated by a simple reduction technique involving either hyperpronation or supination and flexion of the injured arm.3-7

Despite the relative ease of diagnosis and treatment, children with radial head subluxation often wait several hours in a pediatric emergency department for a reduction that takes only a few minutes.8 Such visits have direct health care costs and involve time and stress for the child and their family. While many factors are associated with parental and patient satisfaction in the emergency department, it appears that that early treatment or intervention and shorter waiting times correlate with patient and parent satisfaction.9,10 As well, patient satisfaction appears to be the same or better when emergency department care for minor injuries is provided by nurse practitioners compared to physicians.11-13 Increasingly nurse initiated treatments and the use of medical directives and clinical pathways are becoming a focus in providing health care.14-17 While radial head subluxation treatment is an appropriate area to consider management by emergency department nurses, no studies have examined their role in the management of this common injury. Our study's objective was to examine whether triage nurses, trained in the use of a medical directive that taught recognition and treatment of radial head subluxation, could successfully reduce radial head subluxation at a rate similar to physicians. Given the practical constraints at the time of emergency department triage, this study was designed as a cluster randomized trial where the unit of randomization was a day and the patients on any given day were assigned to the nurse or physician arm for the entire day.

DETAILED DESCRIPTION:
Study design:

We performed an open (i.e. unblinded) non-inferiority, cluster-randomized control trial, to assess whether emergency department triage nurses could, using a medical directive and given specific training, achieve rates of successful reduction of radial head subluxation that were not substantially lower than those of physicians. The Children's Hospital of Eastern Ontario Research Ethics Board approved this study (REB approval number 08-29X). A cluster randomized trial design was used to facilitate the enrollment of patients. The unpredictable acuity and volume of patients presenting to the emergency department triage area made randomization at a patient level unfeasible. Patients were assigned by day of presentation to either nurse or physician treatment. Each day represents a cluster. The anticipated number of children presenting to the emergency department per day with radial head subluxation was less than one, therefore the reduction of power due to clustering was expected to be inconsequential.

Since this study was an assessment of a practice change (medical directive for nurse initiated reduction of presumed radial head subluxation), written, informed consent was deemed unnecessary by the responsible research ethics board. On nurse initiated reduction days verbal consent for the procedure was obtained from caregivers of eligible children prior to the nurse's attempt at reduction. This consent was recorded on the study case report forms.

Study setting and participants:

All children presenting to the emergency department of the Children's Hospital of Eastern Ontario (CHEO) with a presumed diagnosis of radial head subluxation from October 2009 to October 2010 were screened for enrolment. CHEO is a tertiary care pediatric hospital with approximately 55,000 emergency department visits per year at the time of the study. There are about 60 nurses who work in the emergency department, the majority of whom are trained as triage nurses. All triage nurses have a minimum 2 years of experience, attend a compulsory 4-hour orientation course, and complete three 4-hour shifts alongside an experienced triage nurse. Physician coverage includes 26 full-time physicians with specific training in pediatric emergency medicine and 18 part-time staff physicians with other types of training (including general pediatrics, emergency medicine, and family practice), in addition to pediatric emergency fellows, residents, and medical students working under their supervision. Children were eligible for the study if they met the eligibility criteria for the radial head subluxation medical direction (Appendix 1).

Development of medical directive and training of nurses:

A multidisciplinary team developed a medical directive according to our institutional processes. The medical directive permitted triage nurses to attempt a reduction for children presenting with signs and symptoms compatible with radial head subluxation. Children were eligible for the medical directive if they met the following criteria: (1) up to and including 6 years of age, (2) physical exam consistent with radial head subluxation which included not using the affected limb, holding the elbow in extension or slight flexion, forearm in hyperpronation, and distressed only on elbow movement, and (3) injury within preceding 12 hours. Children were excluded from the directive if they had any of the following: (1) an unknown mechanism of injury, (2) deformity of clavicle or arm, (3) swelling of elbow or wrist, (4) significant tenderness on palpation of arm, (5) metabolic bone disease (such as osteogenesis imperfecta), (6) neuromuscular disorder that excluded adequate assessment (such as cerebral palsy), and (7) any concern for abuse or neglect.

A multimodal training initiative was used to educate nurses on the medical directive. This included a short instructional video featuring reduction techniques, a didactic presentation on the physiology and presentation of radial head subluxation, and a hands-on, one hour training session provided by either a study investigator or the study coordinator (a nurse). Training involved instruction on both of the common reduction methods, namely hyperpronation and supination-flexion.4-7 The triage nurses were not allowed to initiate reductions until all training components completed. The medical directive instructed nurses to first use the hyperpronation reduction technique and then the supination-flexion technique, given evidence that hyperpronation may be more successful.18

Study protocol:

A computer-generated randomization calendar schedule was prepared in advance, by the study statistician, for the entire patient recruitment period. The statistician had no role in the recruitment of patients and the investigators were not aware of the schedule in advance. The sequence was composed of randomly permuted blocks with block size of eight. Since the emergency department census can vary daily and seasonally, the use of permuted-block randomization ensured an approximate balance of nurse-initiated and physician-initiated treatment days through the study. The sequence was kept concealed until the beginning of each calendar week, when the sequence for that week was revealed and posted at the throughout the department. The weekly calendar indicated whether the given day was a "nurse-initiated" or "physician-initiated" day.

To ensure comparability of groups, only children who met the criteria for probable radial head subluxation according to the medical directive were eligible for the study on both nurse-initiated and physician-initiated treatment days. Children who, by history, appeared to have radial head subluxation, but had a spontaneous reduction of this injury prior to assessment by the randomized care provider were not included in the study.

On nurse initiated days, children with presumed radial head subluxation were identified by the triage nurses. Once a patient was identified by the triage nurse as having presumed radial head subluxation, the patient's age, sex, arm injured and time and mechanism of injury were prospectively collected using a standardized data form. The triage nurse, with the parent's verbal consent, then attempted reduction, first using the hyperpronation method.4-7 If the child did not begin using their arm normally within 10 minutes of this attempt, a second reduction was attempted via the supination-flexion method.4-7 If at this time point the child still did not have normal arm usage they were placed in the queue to see the emergency department physician as per their triage time and the Pediatric Canadian Triage and Acuity Scale category (pedsCTAS).19 If the reduction was successful (i.e.: child using arm normally) the triage nurse recorded the time of normal arm usage on the standardized data form and an emergency department physician was asked to confirm normal functioning prior to discharge. If the family did not provide verbal consent for the nurse to attempt reduction, the child was placed in the queue to see a physician as per their triage time and triage category.

On physician assigned days, patients with presumed radial head subluxation were typically identified by the triage nurse, who would then place a standardized study data form with the patient's chart, but patients could also be identified by the treating physician. On physician treatment days, children were placed in the queue to see the emergency physician by their triage time and pedsCTAS category. Patients were seen via the usual emergency department practice by either a trainee (medical student, resident, fellow) or staff and treated as per their usual standards. We did not standardize the type or order of reduction manoeuvre for the physician-initiated treatment group. The treating physician was asked to record the time of normal arm usage and reduction method used.

Data was abstracted from the emergency department records of all enrolled children by the study coordinator related to final diagnosis, discharge time, follow-up recommendations, and investigations ordered (such as x-rays) and their results. The study coordinator also completed a daily review of all emergency department charts to determine how many children had a final diagnosis of radial head subluxation during the study, how many of these were enrolled, and of those not enrolled, how many met the medical directive eligibility criteria (based on details documented on the triage document, nursing notes, and physician notes).

ELIGIBILITY:
Inclusion Criteria:

* Age up to 6 years
* Physical exam consistent with RHS which includes not using the affected limb, holding the elbow in extension or slight flexion, forearm in pronation, and patient is distressed only on elbow movement
* Injury within preceding 12 hours

Exclusion Criteria:

* Deformity of clavicle or arm
* Swelling of elbow or wrist
* Significant tenderness on palpation of arm
* Metabolic bone disease (i.e. osteogenesis imperfecta)
* Neuromuscular disorder that excludes adequate assessment (i.e. severe cerebral palsy)

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 245 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Dixon, MD, Principal Investigator — University of Alberta; Amy Plint, MD, Study Director — University of Ottawa; Martin Osmond, MD, Study Director — University of Ottawa; Nick Barrowman, PhD, Study Director — University of Ottawa
Locations (1):
- Childrens Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Schutzman SA, Teach S. Upper-extremity impairment in young children. Ann Emerg Med. 1995 Oct;26(4):474-9. doi: 10.1016/s0196-0644(95)70117-6. PMID 7574131
- [Background] Salter RB, Zaltz C. Anatomic investigations of the mechanism of injury and pathologic anatomy of "pulled elbow" in young children. Clin Orthop Relat Res. 1971;77:134-43. No abstract available. PMID 5140442
- [Background] Quan L, Marcuse EK. The epidemiology and treatment of radial head subluxation. Am J Dis Child. 1985 Dec;139(12):1194-7. doi: 10.1001/archpedi.1985.02140140028018. PMID 4061421
- [Background] Teach SJ, Schutzman SA. Prospective study of recurrent radial head subluxation. Arch Pediatr Adolesc Med. 1996 Feb;150(2):164-6. doi: 10.1001/archpedi.1996.02170270046006. PMID 8556120
- [Background] Jongschaap HC, Youngson GG, Beattie TF. The epidemiology of radial head subluxation ('pulled elbow') in the Aberdeen city area. Health Bull (Edinb). 1990 Mar;48(2):58-61. PMID 2332335
- [Background] Macias CG, Bothner J, Wiebe R. A comparison of supination/flexion to hyperpronation in the reduction of radial head subluxations. Pediatrics. 1998 Jul;102(1):e10. doi: 10.1542/peds.102.1.e10. PMID 9651462
- [Background] Schunk JE. Radial head subluxation: epidemiology and treatment of 87 episodes. Ann Emerg Med. 1990 Sep;19(9):1019-23. doi: 10.1016/s0196-0644(05)82567-3. PMID 2393168
- [Background] McDonald J, Whitelaw C, Goldsmith LJ. Radial head subluxation: comparing two methods of reduction. Acad Emerg Med. 1999 Jul;6(7):715-8. doi: 10.1111/j.1553-2712.1999.tb00440.x. PMID 10433531
- [Background] Taha AM. The treatment of pulled elbow: a prospective randomized study. Arch Orthop Trauma Surg. 2000;120(5-6):336-7. doi: 10.1007/s004020050477. PMID 10853908
- [Background] Toupin P, Osmond MH, Correll R, Plint A. Radial head subluxation: how long do children wait in the emergency department before reduction? CJEM. 2007 Sep;9(5):333-7. PMID 17935648
- [Background] Bursch B, Beezy J, Shaw R. Emergency department satisfaction: what matters most? Ann Emerg Med. 1993 Mar;22(3):586-91. doi: 10.1016/s0196-0644(05)81947-x. PMID 8442550
- [Background] Sacchetti A, Ramoska EE, Glascow C. Nonclassic history in children with radial head subluxations. J Emerg Med. 1990 Mar-Apr;8(2):151-3. doi: 10.1016/0736-4679(90)90224-j. PMID 2362116
- [Background] Choung W, Heinrich SD. Acute annular ligament interposition into the radiocapitellar joint in children (nursemaid's elbow). J Pediatr Orthop. 1995 Jul-Aug;15(4):454-6. doi: 10.1097/01241398-199507000-00008. PMID 7560033
- [Background] Illingworth CM. Pulled elbow: a study of 100 patients. Br Med J. 1975 Jun 21;2(5972):672-4. doi: 10.1136/bmj.2.5972.672. PMID 1139174
- [Background] Green DA, Linares MY, Garcia Pena BM, Greenberg B, Baker RL. Randomized comparison of pain perception during radial head subluxation reduction using supination-flexion or forced pronation. Pediatr Emerg Care. 2006 Apr;22(4):235-8. doi: 10.1097/01.pec.0000210172.17892.a1. PMID 16651912
- [Background] Macias CG, Wiebe R, Bothner J. History and radiographic findings associated with clinically suspected radial head subluxations. Pediatr Emerg Care. 2000 Feb;16(1):22-5. doi: 10.1097/00006565-200002000-00007. PMID 10698138
- [Background] Kaplan RE, Lillis KA. Recurrent nursemaid's elbow (annular ligament displacement) treatment via telephone. Pediatrics. 2002 Jul;110(1 Pt 1):171-4. doi: 10.1542/peds.110.1.171. PMID 12093966
- [Background] Fry M, Holdgate A. Nurse-initiated intravenous morphine in the emergency department: efficacy, rate of adverse events and impact on time to analgesia. Emerg Med (Fremantle). 2002 Sep;14(3):249-54. doi: 10.1046/j.1442-2026.2002.00339.x. PMID 12487041
- [Background] Klassen TP, Ropp LJ, Sutcliffe T, Blouin R, Dulberg C, Raman S, Li MM. A randomized, controlled trial of radiograph ordering for extremity trauma in a pediatric emergency department. Ann Emerg Med. 1993 Oct;22(10):1524-9. doi: 10.1016/s0196-0644(05)81252-1. PMID 8214829
- [Background] Tambimuttu J, Hawley R, Marshall A. Nurse-initiated x-ray of isolated limb fractures in the emergency department: research outcomes and future directions. Aust Crit Care. 2002 Aug;15(3):119-22. doi: 10.1016/s1036-7314(02)80052-2. PMID 12371379
- [Background] Wilmshurst P, Purchase A, Webb C, Jowett C, Quinn T. Improving door to needle times with nurse initiated thrombolysis. Heart. 2000 Sep;84(3):262-6. doi: 10.1136/heart.84.3.262. PMID 10956286
- [Background] Salt P, Clancy M. Implementation of the Ottawa Ankle Rules by nurses working in an accident and emergency department. J Accid Emerg Med. 1997 Nov;14(6):363-5. doi: 10.1136/emj.14.6.363. PMID 9413774
- [Background] Cooper MA, Lindsay GM, Kinn S, Swann IJ. Evaluating Emergency Nurse Practitioner services: a randomized controlled trial. J Adv Nurs. 2002 Dec;40(6):721-30. doi: 10.1046/j.1365-2648.2002.02431.x. PMID 12473052
- [Background] Rhee KJ, Dermyer AL. Patient satisfaction with a nurse practitioner in a university emergency service. Ann Emerg Med. 1995 Aug;26(2):130-2. doi: 10.1016/s0196-0644(95)70141-9. PMID 7618773
- [Background] Moser MS, Abu-Laban RB, van Beek CA. Attitude of emergency department patients with minor problems to being treated by a nurse practitioner. CJEM. 2004 Jul;6(4):246-52. doi: 10.1017/s1481803500009209. PMID 17382000
- [Background] Magaret ND, Clark TA, Warden CR, Magnusson AR, Hedges JR. Patient satisfaction in the emergency department--a survey of pediatric patients and their parents. Acad Emerg Med. 2002 Dec;9(12):1379-88. doi: 10.1197/aemj.9.12.1379. PMID 12460841
- [Background] Moher D, Schulz KF, Altman D; CONSORT Group (Consolidated Standards of Reporting Trials). The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomized trials. JAMA. 2001 Apr 18;285(15):1987-91. doi: 10.1001/jama.285.15.1987. PMID 11308435
- [Background] Amir D, Frankl U, Pogrund H. Pulled elbow and hypermobility of joints. Clin Orthop Relat Res. 1990 Aug;(257):94-9. PMID 2379380
- [Background] Snyder HS. Radiographic changes with radial head subluxation in children. J Emerg Med. 1990 May-Jun;8(3):265-9. doi: 10.1016/0736-4679(90)90003-e. PMID 2373834
- [Background] Newcombe RG. Interval estimation for the difference between independent proportions: comparison of eleven methods. Stat Med. 1998 Apr 30;17(8):873-90. doi: 10.1002/(sici)1097-0258(19980430)17:83.0.co;2-i. PMID 9595617
- [Background] Donner A, Donald A. The statistical analysis of multiple binary measurements. J Clin Epidemiol. 1988;41(9):899-905. doi: 10.1016/0895-4356(88)90107-2. PMID 3183697
- [Background] Kerry SM, Bland JM. Analysis of a trial randomised in clusters. BMJ. 1998 Jan 3;316(7124):54. doi: 10.1136/bmj.316.7124.54. No abstract available. PMID 9451271
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] Plint AC, Johnson DW, Wiebe N, Bulloch B, Pusic M, Joubert G, Pianosi P, Turner T, Thompson G, Klassen TP. Practice variation among pediatric emergency departments in the treatment of bronchiolitis. Acad Emerg Med. 2004 Apr;11(4):353-60. doi: 10.1197/j.aem.2003.12.003. PMID 15064208
- [Background] Bjornson CL, Klassen TP, Williamson J, Brant R, Mitton C, Plint A, Bulloch B, Evered L, Johnson DW; Pediatric Emergency Research Canada Network. A randomized trial of a single dose of oral dexamethasone for mild croup. N Engl J Med. 2004 Sep 23;351(13):1306-13. doi: 10.1056/NEJMoa033534. PMID 15385657
- [Background] Plint AC, Perry JJ, Correll R, Gaboury I, Lawton L. A randomized, controlled trial of removable splinting versus casting for wrist buckle fractures in children. Pediatrics. 2006 Mar;117(3):691-7. doi: 10.1542/peds.2005-0801. PMID 16510648
- [Background] Casarett D, Karlawish JH, Sugarman J. Determining when quality improvement initiatives should be considered research: proposed criteria and potential implications. JAMA. 2000 May 3;283(17):2275-80. doi: 10.1001/jama.283.17.2275. PMID 10807388
- [Background] Lynn J, Baily MA, Bottrell M, Jennings B, Levine RJ, Davidoff F, Casarett D, Corrigan J, Fox E, Wynia MK, Agich GJ, O'Kane M, Speroff T, Schyve P, Batalden P, Tunis S, Berlinger N, Cronenwett L, Fitzmaurice JM, Dubler NN, James B. The ethics of using quality improvement methods in health care. Ann Intern Med. 2007 May 1;146(9):666-73. doi: 10.7326/0003-4819-146-9-200705010-00155. Epub 2007 Apr 16. PMID 17438310
- [Derived] Dixon A, Clarkin C, Barrowman N, Correll R, Osmond MH, Plint AC. Reduction of radial-head subluxation in children by triage nurses in the emergency department: a cluster-randomized controlled trial. CMAJ. 2014 Jun 10;186(9):E317-23. doi: 10.1503/cmaj.131101. Epub 2014 Mar 24. PMID 24664649

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 Patients in the physician group were incorrectly reduced by the triage nurse 21 patients in the nurse group either had no study form or the nurse did not attempt reduction
Period: Overall Study
Arm/Group | Nurse Reduction | Physician Reduction
Started | 145 | 123
Completed | 124 | 121
Not Completed | 21 | 2
Not completed — Protocol Violation | 21 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nurse Reduction | Physician Reduction | Total
Number analyzed (Participants) | 124 | 121 | 245
Age, Continuous [Mean (Standard Deviation); unit: Years] | 2.4 (1.0) | 2.2 (1.1) | 2.3 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 68 | 148
  Male | 44 | 53 | 97
Region of Enrollment [Number; unit: participants]
  Canada | 124 | 121 | 245
Time from injury [Median (Inter-Quartile Range); unit: Minutes] | 88 [45 to 153] | 103 [64 to 199] | 92 [54 to 173]
Number of patient with injury from pull mechanism [Number; unit: participants] | 118 | 92 | 210
Number of patients with injury from fall mechanism [Number; unit: participants] | 5 | 19 | 24
Number of patient with injury from other mechanisms [Number; unit: participants] | 1 | 10 | 11

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Successful Reduction of Radial Head Subluxation by Nurse, Compared With Physician Controls
Time Frame: 10-15 minutes post reduction attempt
Measure: Number; unit: percentage of patients reduced
Arm/Group | Nurse Reduction | Physician Reduction
Number analyzed (Participants) | 124 | 121
percentage of patients reduced | 84.7 | 96.7

2. Secondary Outcome: Time to Discharge From ED (Minutes)
Time Frame: End of enrollment
Population: 2 missing data point in the physician group
Measure: Median (Full Range); unit: minutes
Arm/Group | Nurse Reduction | Physician Reduction
Number analyzed (Participants) | 124 | 119
minutes | 50 [32 to 82] | 105 [63 to 150]

3. Secondary Outcome: Proportion of Patients With Presentation Compatible With RHS, Have Reduction Attempted, Who Are Subsequently Diagnosed With Fracture.
Time Frame: Every 3 months during enrollment
Measure: Number; unit: participants
Arm/Group | Nurse Reduction | Physician Reduction
Number analyzed (Participants) | 124 | 121
participants | 1 | 0

4. Secondary Outcome: Proportion of Patients With RHS Not Identified by Nurse Pathway.
Time Frame: End of enrollment
Measure: Number; unit: participants
Arm/Group | Nurse Reduction
Number analyzed (Participants) | 145
participants | 21

ADVERSE EVENTS:
Groups:
- Physician Reduction: Patients randomized to reduction by physician
  Physicians were free to use the reduction method of their choice
Arm/Group | Nurse Reduction | Physician Reduction
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/123
Other Adverse Events (participants affected / at risk) | 1/145 | 0/123
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nurse Reduction (N=145) | Physician Reduction (N=123)
Reduction attempted, subsequent fracture diagnosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — 1 patient in nurse group had a reduction attempted and was later found to have a type 1 supracondylar fracture. This healed well with good recovery of function. There was unneccesary pain from the reduction attempt

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No